CLINICAL TRIAL: NCT02432508
Title: Efficacy of Laser Acupuncture on Pruritus in Patients With Chronic Kidney Disease Undergoing Hemodialysis: A Multiple Centers, Randomized, Assessor- and Participant-blind, Controlled, Cross-over Clinical Trial
Brief Title: Efficacy of Laser Acupuncture on Pruritus in Patients With Chronic Kidney Disease Undergoing Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A-3-2-A/CMUH103-REC2-112
Record Dates: First submitted 2015-01-18; First posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Pruritus; Kidney Failure, Chronic
Keywords: acupuncture; laser; uremic pruritus; randomized clinical trial
MeSH Terms: conditions — Pruritus; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laser acupuncture (Active Comparator): One hundreds of hemodialysis patients include and give intervention with laser acupuncture (50mW) for 4 weeks. After 4 weeks of wash out period, these patients cross over to shame laser acupuncture treatment (5mW).
  Interventions: Device: Laser acupuncture (Olympic); Device: Sham Laser acupuncture (Olympic)
- sham laser acupuncture (Sham Comparator): One hundreds of hemodialysis patients include and give intervention with sham laser acupuncture (5mW) for 4 weeks. After 4 weeks of wash out period, these patients cross over to laser acupuncture treatment (50mW).
  Interventions: Device: Laser acupuncture (Olympic); Device: Sham Laser acupuncture (Olympic)

INTERVENTIONS:
Device: Laser acupuncture (Olympic) — Physiolaser Olympic laser acupuncture device (50mW, 655nm)
Device: Sham Laser acupuncture (Olympic) — Physiolaser Olympic laser acupuncture device (Low dose of laser energy: 5mW, 655nm)

SUMMARY:
Uremic pruritus is a clinically significant symptom which imposes heavy impact on the quality of life of patients with chronic kidney disease undergoing hemodialysis. In order to investigate the clinical efficacy and mechanism, the investigators designed a multiple centers, randomized, assessor- and participant-blind, controlled, cross-over clinical trial. This trial will be conducted at Taichung branch, Feng-yuan branch and the Eastern branch of CMUH.

DETAILED DESCRIPTION:
We plan to enroll 200 volunteer patients with uremic pruritus. After the waiting period (as the waiting list group), you will be randomized to laser acupuncture and sham laser acupuncture group. Each group will include 100 patients and given intervention according to their hemodialysis frequency, i.e., BIW or TIW. The intervention will then be crossed over to the other one after 4 week of wash-our period. Outcome measurement includes questionnaires, biochemistry analysis, instrumental analysis and medication score.

ELIGIBILITY:
Inclusion Criteria:

* Age>20y/o, ESRD patient, pruritus symptoms persist longer than 4 weeks

Exclusion Criteria:

* immunosupression agents use, undergo chemotherapy
* drug abuser
* pregnancy women
* patient with psychiological disorder
* arrhythemia, pacemaker device use
* local skin infection over laser acupuncture site
* patient allergy to laser acupuncture treament

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pruritus Visual Analogue Scale | 20 weeks
  We plan to enroll 200 volunteer patients with uremic pruritus. After the waiting period (4weeks), the patients will be randomized to laser acupuncture and sham laser acupuncture group (4weeks). Each group will include 100 patients and given intervention according to their hemodialysis frequency, i.e., BIW or TIW. The intervention will then be crossed over to the other one after 4 week of wash-our period. Outcome measurement includes questionnaires, biochemistry analysis, instrumental analysis and medication score will perform in the last 4 weeks.
  Pruritus Visual Aaalogue Scale questionnaire will perform on each visit of hemodialysis.

SECONDARY OUTCOMES:
Short-Form-36 Health Survey (SF-36) | 20 weeks
  SF-36 questionnaire will perform in the begin, 4th, 8th, 12th, 16th and 20th week.
Dermatology Life Quality Index (DLQI) | 20 weeks
  DLQI questionnaire will perform in the begin, 4th, 8th, 12th, 16th and 20th week.
The 5-D itch scale | 20 weeks
  The 5-D itch scale will perform in the begin, 4th, 8th, 12th, 16th and 20th week.
The Pittsburgh Sleep Quality Index; PSQI | 20 weeks
  PSQI will perform in the begin, 4th, 8th, 12th, 16th and 20th week.
Beck Depression Inventory, BDI | 20 weeks
  BDI will perform in the begin, 4th, 8th, 12th, 16th and 20th week.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chiz-Tzung, Ph.D., Study Chair — School of Medicine, China Medical University
Locations (1):
- China Medical University Hospital, Taichung, Taichung, Taiwan

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264